CLINICAL TRIAL: NCT05809050
Title: Study of miRNA-155 in Acute Leukemia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Noura Farouk Abdallah, clinical pathology specialist at sohag university, Sohag University
Other Study IDs: Soh-Med-23-03-01MD
Record Dates: First submitted 2023-03-30; First posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-03

CONDITIONS: Acute Leukemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control group: represents the control group ( ITP cases
  Interventions: Diagnostic Test: BM aspirate
- AL group: cases of AcuteLeukemia.
  Interventions: Diagnostic Test: BM aspirate

INTERVENTIONS:
Diagnostic Test: BM aspirate — Bone Marrow aspiration & Examination

SUMMARY:
The leukaemias are a heterogeneous group of blood cancers, Acute leukaemia (AL) is caused by malignant proliferation of blood cells arrested at an immature stage of development, They are very aggressive diseases that run a rapidly fatal course if not promptly diagnosed and appropriately treated. Misdiagnosis is very common with delay in diagnosis and prompt treatment being the causes of high morbidity and mortality in acute leukaemias.

Although with the continuous improvement of clinical and laboratory diagnosis and treatment methods, the prognosis of AML has been significantly improved, but there are still about 70% of patients who cannot survive more than 5 years after diagnosis The activity of miRNAs in tumors is regulated by the same alterations affecting protein-coding genes, such as chromosomal rearrangements, genomic amplifications or deletions or mutations, abnormal transcriptional control, dysregulation of epigenetic changes and defects in the biogenesis machinery A typical chromosomal rearrangement is a chromosomal translocation, especially in hematological malignancies, in which it promotes tumor development and progression by the promoter exchange or by the creation of chimeric genes translated as fusion proteins. In Acute Myeloid Leukemia (AML) patients with myeloid/lymphoid leukemia gene (or mixed-lineage leukemia, MLL) rearrangement, by large-scale genome-wide microarray analysis, it was demonstrated that among 48 selected miRNAs, 47 of them are increased

ELIGIBILITY:
Inclusion Criteria:

* approval to sign an informed written consent, patient with newly diagnosed AL.

Exclusion Criteria:

* Refusal to sign an informed written consent, Cases with Chronic leukemias, Lymphoma or Leukemic phase of lymphoma or patients on chemotherapy.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Group (I): represents the control group ( ITP cases). Group (II): represents the cases of Acute Leukemia.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Detection of miRNA-155 | one year
  Detection of miRNA-155 using real time PCR on bone marrow aspirate samples

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kirtonia A, Pandya G, Sethi G, Pandey AK, Das BC, Garg M. A comprehensive review of genetic alterations and molecular targeted therapies for the implementation of personalized medicine in acute myeloid leukemia. J Mol Med (Berl). 2020 Aug;98(8):1069-1091. doi: 10.1007/s00109-020-01944-5. Epub 2020 Jul 3. PMID 32620999
- [Background] Culp-Hill R, D'Alessandro A, Pietras EM. Extinguishing the Embers: Targeting AML Metabolism. Trends Mol Med. 2021 Apr;27(4):332-344. doi: 10.1016/j.molmed.2020.10.001. Epub 2020 Oct 26. PMID 33121874
- [Background] Dachi RA, Mustapha FG, Mahdi M, Abbas H. Acute Leukaemias in Bauchi State, Northeastern Nigeria: Pattern of Presentations and Clinical Entities. West Afr J Med. 2022 May 27;39(5):497-500. PMID 35633629
- [Background] Lefeivre T, Jones L, Trinquand A, Pinton A, Macintyre E, Laurenti E, Bond J. Immature acute leukaemias: lessons from the haematopoietic roadmap. FEBS J. 2022 Aug;289(15):4355-4370. doi: 10.1111/febs.16030. Epub 2021 Jun 10. PMID 34028982